CLINICAL TRIAL: NCT05235750
Title: Self-affirmation Intervention for People Newly Diagnosed With Advanced Cancer: A Preliminary Efficacy Trial
Brief Title: Self-affirmation Intervention for People Newly Diagnosed With Advanced Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 273876
Record Dates: First submitted 2022-02-01; First posted 2022-02-11 (Actual); Results first posted 2025-03-17 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2024-12

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Writing (Experimental): This is a single-group study with one arm only.
  Interventions: Behavioral: Self-affirmation writing

INTERVENTIONS:
Behavioral: Self-affirmation writing — Writing with a focus on self-affirmation at the time following a diagnosis of an advanced cancer

SUMMARY:
The goal of this clinical trial is to learn if a brief writing intervention works to improve quality of life outcomes in adult patients newly diagnosed with advanced stage cancer.

DETAILED DESCRIPTION:
A diagnosis of cancer may challenge one's former assumptions and beliefs about themselves and the world and potentially compromise quality of life (QoL). The primary aim of the study is to explore the preliminary efficacy of an intervention to protect individuals from the negative psychological impact of the cancer diagnosis. The secondary aim is to test the validity of the Functional Assessment of Chronic Illness Therapy- Spiritual Well-Being 12 item Scale (FACIT-Sp-12), in its current and revised forms. Potential participants will be enrolled from two study sites as per protocol: the Winthrop P. Rockefeller Cancer Institute at the University of Arkansas for Medical Sciences (UAMS) and the Arkansas Hospice respectively, and will be asked to write as guided by the researcher for 4 weeks. Study outcomes will be assessed at baseline, 2-, 6- and 8-weeks post baseline. It is hypothesized that self-affirmation via writing at the time following a diagnosis of an advanced cancer by affirming values or beliefs that are salient to self will help enhance self-esteem, reinforce spiritual well-being, decrease levels of anxiety or depression, and improve QoL.

ELIGIBILITY:
Inclusion Criteria:

* within 8 weeks of being informed of diagnosis (primary or recurrent)
* cancer stage III or IV of a primary solid tumor, or a high-grade hematological malignancy, and
* age 18 years or older

Exclusion Criteria:

* medical condition precluding participation (e.g., too ill or fatigued, acute mental confusion as determined by the treating physician), or
* enrolled in other psychosocial experiments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2022-05-27 (Actual); Primary Completion 2023-07-07 (Actual); Study Completion 2023-07-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mei Bai, Ph.D., Principal Investigator — University of Arkansas
Locations (2):
- United States (2):
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Arkansas Hospice, North Little Rock, Arkansas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bai M, Cella D, Jeon S, Govindarajan R, Birrer MJ. Self-affirmation intervention for patients newly diagnosed with advanced cancer: a preliminary efficacy trial. J Psychosoc Oncol. 2025;43(4):593-615. doi: 10.1080/07347332.2025.2450013. Epub 2025 Jan 15. PMID 39812781

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Writing
Started | 57
Completed | 45
Not Completed | 12

BASELINE CHARACTERISTICS:
Population: Two patients were deceased shortly after enrollment and one was unable to reach again, leaving a total of 54 participants who were able to complete baseline data.
Arm/Group | Writing
Number analyzed (Participants) | 54
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 29
  >=65 years | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.8 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 27
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Caucasian | 41
  Race: African American | 12
  Race: Asian | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: non-Hispanic | 54
  Ethnicity: Hispanic | 0
Education [Count of Participants; unit: Participants]
  Up to 8th grade | 1
  High school | 21
  College | 26
  Graduate school | 5
  Unknown or not reported | 1
Marital status [Count of Participants; unit: Participants]
  single | 7
  married | 31
  divorced | 9
  widowed | 7
Religious affiliation [Count of Participants; unit: Participants]
  None | 10
  Protestant | 17
  Catholic | 3
  Other | 23
  Undisclosed | 1
Time since cancer diagnosis [Mean (Standard Deviation); unit: days] | 46.3 (23.5)
Stage of cancer [Count of Participants; unit: Participants]
  III | 17
  IV | 31
  recurrent | 2
  unstaged | 4
Cancer site [Count of Participants; unit: Participants]
  Gastrointestinal (GI) | 18
  Lung | 13
  Gynecological (GYN) | 10
  Head and neck | 7
  Prostate | 3
  Breast | 2
  Hematological | 1
Preference to talk [Count of Participants; unit: Participants]
  yes | 33
  no | 13
  not sure | 8
Ever wrote a diary in life [Count of Participants; unit: Participants]
  no | 38
  yes | 16
Should one have a religious affiliation to be spiritual? [Count of Participants; unit: Participants]
  no | 37
  yes | 17
Perceived threat from cancer diagnosis [Count of Participants; unit: Participants]
  a great deal threatening | 16
  moderately threatening | 14
  a little threatening | 13
  not or hardly threatening | 11

OUTCOME MEASURES:

1. Primary Outcome: Mean Changes From Baseline in Self-esteem Scores on the Rosenberg Self-esteem Scale (RSES) to Two-, Six-, and Eight Weeks Post Baseline
Description: Changes include raw score changes and standardized mean differences. Scores on the Rosenberg Self-esteem Scale range from 0 to 30, with higher score indicating higher level of self-esteem.
Time Frame: Baseline (T1) as well as 2 weeks (T2), 6 weeks (T3), and 8 weeks post baseline (T4)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Writing
Number analyzed (Participants) | 54
score on a scale
  RSES at T1 | 23.4 (3.8)
  RSES at T2 | 23.5 (4.1)
  RSES at T3 | 23.7 (4.2)
  RSES at T4 | 24.2 (4.7)
Statistical Analysis 1: Comparison: Writing; We analyzed short- (at 6 weeks post-baseline or T3) and longer-term differences (at 8 weeks post-baseline or T4) for the RSES, expecting a larger size of differences at T3. The short-term difference [(T3-T2)-(T2-T1)] represents differences between post-intervention change (T3-T2) and pre-intervention change (T2-T1). Longer-term difference [(T4-T2)-(T2-T1)] represents differences between 2 weeks post-intervention change (T4-T2) and pre-intervention change (T2-T1); Test type: Other; p = .83, Mixed Models Analysis — The above p value refers to the difference between post-intervention change and pre-intervention change (or [(T3-T2)-(T2-T1)]) for RSES; Mean Difference (Net) = 0.2 — The above value represents net difference between post-intervention change and pre-intervention change (or [(T3-T2)-(T2-T1)]) for RSES
Statistical Analysis 2: Comparison: Writing; Test type: Other; p = .91, Mixed Models Analysis — The above p value refers to the difference between 2 weeks post-intervention change and pre-intervention change (or [(T4-T2)-(T2-T1)]) for RSES; Mean Difference (Net) = -0.2 — The above value represents net difference between 2 weeks post-intervention change and pre-intervention change (or [(T4-T2)-(T2-T1)]) for RSES

2. Primary Outcome: Mean Changes From Baseline in Quality of Life (QoL) Scores on the Functional Assessment of Cancer Therapy-General (FACT-G) to Two-, Six-, and Eight Weeks Post Baseline
Description: Changes include raw score changes and standardized mean differences. Scores on the Functional Assessment of Cancer Therapy-General (FACT-G) range from 0 to 108, with higher score indicating higher level of quality of life. Each subscale ranging from 0 to 28, with higher score indicating higher level of quality of life. The raw scores of overall QoL (total FACT-G), four composite domains (physical well-being, PWB; social/family well-being, SWB; emotional well-being, EWB; functional well-being, FWB), global QoL (item Gf7 "I am content with the quality of my life right now") and one item pertinent to this study (Ge6 "I worry that my condition will get worse") were presented below.
Time Frame: Baseline (T1) as well as 2 weeks (T2), 6 weeks (T3), and 8 weeks post baseline (T4)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Writing
Number analyzed (Participants) | 54
score on a scale
  FACT-G (total score) at T1 | 78.7 (15.2)
  FACT-G (total score) at T2 | 80.7 (16.3)
  FACT-G (total score) at T3 | 80.7 (14.9)
  FACT-G (total score) at T4 | 81.2 (17.0)
  PWB at T1 | 20.6 (4.8)
  PWB at T2 | 19.4 (6.0)
  PWB at T3 | 19.3 (5.3)
  PWB at T4 | 19.5 (5.7)
  SWB at T1 | 22.7 (4.4)
  SWB at T2 | 24.1 (4.3)
  SWB at T3 | 23.5 (4.2)
  SWB at T4 | 23.6 (4.4)
  EWB at T1 | 18.6 (3.9)
  EWB at T2 | 19.1 (4.4)
  EWB at T3 | 19.3 (4.5)
  EWB at T4 | 19.5 (4.5)
  FWB at T1 | 16.8 (6.8)
  FWB at T2 | 18.1 (6.3)
  FWB at T3 | 18.7 (5.7)
  FWB at T4 | 18.5 (6.2)
  Gf7 at T1 | 2.4 (1.3)
  Gf7 at T2 | 2.6 (1.2)
  Gf7 at T3 | 2.7 (1.3)
  Gf7 at T4 | 2.6 (1.2)
  Ge6 at T1 | 2.8 (1.1)
  Ge6 at T2 | 2.8 (1.2)
  Ge6 at T3 | 3.0 (1.2)
  Ge6 at T4 | 3.0 (1.1)
Statistical Analysis 1: Comparison: Writing; We analyzed short- (at 6 weeks post-baseline, T3) and longer-term differences (at 8 weeks post-baseline, T4) for the FACT-G at scale, factor and item levels expecting a larger size of differences at T3. The short-term difference [(T3-T2)-(T2-T1)] represents differences between post-intervention change (T3-T2) and pre-intervention change (T2-T1). Longer-term difference [(T4-T2)-(T2-T1)] represents differences between 2 weeks post-intervention change (T4-T2) and pre-intervention change (T2-T1); Test type: Other; p = .45, Mixed Models Analysis — The above p value refers to the difference between post-intervention change and pre-intervention change (or [(T3-T2)-(T2-T1)]) for the total FACT-G; Mean Difference (Net) = -2.1 — The above value represents net difference between post-intervention change and pre-intervention change (or [(T3-T2)-(T2-T1)]) for the total FACT-G
Statistical Analysis 2: Comparison: Writing; Test type: Other; p = .29, Mixed Models Analysis — The above p value refers to the difference between 2 weeks post-intervention change and pre-intervention change (or [(T4-T2)-(T2-T1)]) for the total FACT-G; Mean Difference (Net) = -3.3 — The above value represents net difference between 2 weeks post-intervention change and pre-intervention change (or [(T4-T2)-(T2-T1)]) for the total FACT-G
Statistical Analysis 3: Comparison: Writing; Test type: Other; p = .46, Mixed Models Analysis — The above p value refers to the difference between post-intervention change and pre-intervention change (or [(T3-T2)-(T2-T1)]) for physical well-being (PWB) as measured by the FACT-G; Mean Difference (Net) = 0.8 — The above value represents net difference between post-intervention change and pre-intervention change (or [(T3-T2)-(T2-T1)]) for physical well-being (PWB) as measured by the FACT-G
Statistical Analysis 4: Comparison: Writing; Test type: Other; p = .79, Mixed Models Analysis — The above p value refers to the difference between 2 weeks post-intervention change and pre-intervention change (or [(T4-T2)-(T2-T1)]) for physical well-being (PWB) as measured by the FACT-G; Mean Difference (Net) = 0.2 — The above value represents net difference between 2 weeks post-intervention change and pre-intervention change (or [(T4-T2)-(T2-T1)]) for physical well-being (PWB) as measured by the FACT-G
Statistical Analysis 5: Comparison: Writing; Test type: Other; p = .05, Mixed Models Analysis — The above p value refers to the difference between post-intervention change and pre-intervention change (or [(T3-T2)-(T2-T1)]) for social/family well-being (SWB) as measured by the FACT-G; Mean Difference (Net) = -2.1 — The above value represents net difference between post-intervention change and pre-intervention change (or [(T3-T2)-(T2-T1)]) for social/family well-being (SWB) as measured by the FACT-G
Statistical Analysis 6: Comparison: Writing; Test type: Other; p = .03, Mixed Models Analysis — The above p value refers to the difference between 2 weeks post-intervention change and pre-intervention change (or [(T4-T2)-(T2-T1)]) for social/family well-being (SWB) as measured by the FACT-G; Mean Difference (Net) = -2.4 — The above value represents net difference between 2 weeks post-intervention change and pre-intervention change (or [(T4-T2)-(T2-T1)]) for social/family well-being (SWB) as measured by the FACT-G
Statistical Analysis 7: Comparison: Writing; Test type: Other; p = .82, Mixed Models Analysis — The above p value refers to the difference between post-intervention change and pre-intervention change (or [(T3-T2)-(T2-T1)]) for emotional well-being (EWB) as measured by the FACT-G; Mean Difference (Net) = -0.2 — The above value represents net difference between post-intervention change and pre-intervention change (or [(T3-T2)-(T2-T1)]) for emotional well-being (EWB) as measured by the FACT-G
Statistical Analysis 8: Comparison: Writing; Test type: Other; p = .58, Mixed Models Analysis — The above p value refers to the difference between 2 weeks post-intervention change and pre-intervention change (or [(T4-T2)-(T2-T1)]) for emotional well-being (EWB) as measured by the FACT-G; Mean Difference (Net) = -0.5 — The above value represents net difference between 2 weeks post-intervention change and pre-intervention change (or [(T4-T2)-(T2-T1)]) for emotional well-being (EWB) as measured by the FACT-G
Statistical Analysis 9: Comparison: Writing; Test type: Other; p = .56, Mixed Models Analysis — The above p value refers to the difference between post-intervention change and pre-intervention change (or [(T3-T2)-(T2-T1)]) for functional well-being (FWB) as measured by the FACT-G; Mean Difference (Net) = -0.8 — The above value represents net difference between post-intervention change and pre-intervention change (or [(T3-T2)-(T2-T1)]) for functional well-being (FWB) as measured by the FACT-G
Statistical Analysis 10: Comparison: Writing; Test type: Other; p = .58, Mixed Models Analysis — The above p value refers to the difference between 2 weeks post-intervention change and pre-intervention change (or [(T4-T2)-(T2-T1)]) for functional well-being (FWB) as measured by the FACT-G; Mean Difference (Net) = -0.7 — The above value represents net difference between 2 weeks post-intervention change and pre-intervention change (or [(T4-T2)-(T2-T1)]) for functional well-being (FWB) as measured by the FACT-G
Statistical Analysis 11: Comparison: Writing; Test type: Other; p = .58, Mixed Models Analysis — The above p value refers to the difference between post-intervention change and pre-intervention change (or [(T3-T2)-(T2-T1)]) for Global QoL (item G7 "I am content with the quality of my life right now") as measured by the FACT-G; Mean Difference (Net) = -0.2 — The above value represents net difference between post-intervention change and pre-intervention change (or [(T3-T2)-(T2-T1)]) for Global QoL (item G7 "I am content with the quality of my life right now") as measured by the FACT-G
Statistical Analysis 12: Comparison: Writing; Test type: Other; p = .34, Mixed Models Analysis — The above p value refers to the difference between 2 weeks post-intervention change and pre-intervention change (or [(T4-T2)-(T2-T1)] for Global QoL (item G7 "I am content with the quality of my life right now") as measured by the FACT-G; Mean Difference (Net) = -0.3 — The above value represents net difference between 2 weeks post-intervention change and pre-intervention change (or [(T4-T2)-(T2-T1)]) for Global QoL (item G7 "I am content with the quality of my life right now") as measured by the FACT-G
Statistical Analysis 13: Comparison: Writing; Test type: Other; p = .27, Mixed Models Analysis — The above p value refers to the difference between post-intervention change and pre-intervention change (or [(T3-T2)-(T2-T1)]) for item Ge6 "I worry that my condition will get worse" as measured by the FACT-G; Mean Difference (Net) = 0.4 — The above value represents net difference between post-intervention change and pre-intervention change (or [(T3-T2)-(T2-T1)]) for item Ge6 "I worry that my condition will get worse" as measured by the FACT-G
Statistical Analysis 14: Comparison: Writing; Test type: Other; p = .62, Mixed Models Analysis — The above p value refers to the difference between 2 weeks post-intervention change and pre-intervention change (or [(T4-T2)-(T2-T1)]) for item Ge6 "I worry that my condition will get worse" as measured by the FACT-G; Mean Difference (Net) = 0 — The above value represents net difference between 2 weeks post-intervention change and pre-intervention change (or [(T4-T2)-(T2-T1)]) for item Ge6 "I worry that my condition will get worse" as measured by the FACT-G

3. Secondary Outcome: Mean Changes From Baseline in Spiritual Well-Being Scores on the Functional Assessment of Chronic Illness Therapy-Spiritual Well-Being 12 Item Scale (FACIT-Sp-12) to Two-, Six-, and Eight Weeks Post Baseline
Description: Changes include raw score changes and standardized mean differences. The FACIT-Sp-12 scale measures an individual's level of spiritual well-being, specifically assessing their sense of meaning, peace, and faith in life, with higher scores indicating a better level of spiritual well-being and lower scores a worse level of spiritual well-being. It consists of 12 items rated on a 5-point Likert scale (0 = Not at all to 4 = Very much). The FACIT-Sp-12 Scale consists of 2 sub-scales Meaning/Peace (M/P) with a range of 0-32, and Faith ranging from 1-16. Possible overall spiritual well-being or FACIT-Sp-12 (total) range from 0 to 48. The revised Faith subscale as well as the revised FACIT-Sp-12 scale have the same scale range of the original measures.
Time Frame: Baseline (T1) as well as 2 weeks (T2), 6 weeks (T3), and 8 weeks post baseline (T4)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Writing
Number analyzed (Participants) | 54
score on a scale
  FACIT-Sp-12 (total) at T1 | 39.5 (8.2)
  FACIT-Sp-12 (total) at T2 | 40.5 (6.8)
  FACIT-Sp-12 (total) at T3 | 41.0 (7.0)
  FACIT-Sp-12 (total) at T4 | 40.0 (8.0)
  M/P at T1 | 26.6 (5.3)
  M/P at T2 | 27.2 (4.3)
  M/P at T3 | 26.9 (5.0)
  M/P at T4 | 26.8 (5.7)
  Faith at T1 | 12.9 (3.9)
  Faith at T2 | 13.2 (3.5)
  Faith at T3 | 14.1 (3.1)
  Faith at T4 | 13.2 (3.6)
  Faith (revised) at T1 | 13.2 (3.5)
  Faith (revised) at T2 | 13.7 (2.9)
  Faith (revised) at T3 | 14.1 (2.9)
  Faith (revised) at T4 | 13.5 (3.4)
  FACIT-Sp-12 total (revised) at T1 | 39.8 (7.7)
  FACIT-Sp-12 total (revised) at T2 | 40.9 (6.6)
  FACIT-Sp-12 total (revised) at T3 | 40.9 (6.9)
  FACIT-Sp-12 total (revised) at T4 | 39.8 (8.3)
Statistical Analysis 1: Comparison: Writing; We analyzed short- (at 6 weeks post-baseline, T3) and longer-term differences (at 8 weeks post-baseline, T4) for the FACIT-Sp-12 at scale and factor levels, expecting a larger size of differences at T3. The short-term difference [(T3-T2)-(T2-T1)] represents differences between post-intervention change (T3-T2) and pre-intervention change (T2-T1). Longer-term difference [(T4-T2)-(T2-T1)] represents differences between 2 weeks post-intervention change (T4-T2) and pre-intervention change (T2-T1); Test type: Other; p = .76, Mixed Models Analysis — The above p value refers to the difference between post-intervention change and pre-intervention change (or [(T3-T2)-(T2-T1)]) for the total FACIT-Sp-12; Mean Difference (Net) = -0.6 — The above value represents net difference between post-intervention change and pre-intervention change (or [(T3-T2)-(T2-T1)]) for the total FACIT-Sp-12
Statistical Analysis 2: Comparison: Writing; Test type: Other; p = .19, Mixed Models Analysis — The above p value refers to the difference between 2 weeks post-intervention change and pre-intervention change (or [(T4-T2)-(T2-T1)]) for the total FACIT-Sp-12; Mean Difference (Net) = -2.1 — The above value represents net difference between 2 weeks post-intervention change and pre-intervention change (or [(T4-T2)-(T2-T1)]) for the total FACIT-Sp-12
Statistical Analysis 3: Comparison: Writing; Test type: Other; p = .35, Mixed Models Analysis — The above p value refers to the difference between post-intervention change and pre-intervention change (or [(T3-T2)-(T2-T1)]) for the Meaning/Peace factor (M/P) as measured by the FACIT-Sp-12; Mean Difference (Net) = -1.0 — The above value represents net difference between post-intervention change and pre-intervention change (or [(T3-T2)-(T2-T1)]) for the Meaning/Peace factor (M/P) as measured by the FACIT-Sp-12
Statistical Analysis 4: Comparison: Writing; Test type: Other; p = .99, Mixed Models Analysis — The above p value refers to the difference between 2 weeks post-intervention change and pre-intervention change (or [(T4-T2)-(T2-T1)]) for the Meaning/Peace factor (M/P) as measured by the FACIT-Sp-12; Mean Difference (Net) = -1.9 — The above value represents net difference between 2 weeks post-intervention change and pre-intervention change (or [(T4-T2)-(T2-T1)]) for the Meaning/Peace factor (M/P) as measured by the FACIT-Sp-12
Statistical Analysis 5: Comparison: Writing; Test type: Other; p = .46, Mixed Models Analysis — The above p value refers to the difference between post-intervention change and pre-intervention change (or [(T3-T2)-(T2-T1)]) for the Faith factor of the FACIT-Sp-12; Mean Difference (Net) = 0.4 — The above value represents net difference between post-intervention change and pre-intervention change (or [(T3-T2)-(T2-T1)]) for the Faith factor of the FACIT-Sp-12
Statistical Analysis 6: Comparison: Writing; Test type: Other; p = .24, Mixed Models Analysis — The above p value refers to the difference between 2 weeks post-intervention change and pre-intervention change (or [(T4-T2)-(T2-T1)]) for the Faith factor of the FACIT-Sp-12; Mean Difference (Net) = -0.7 — The above value represents net difference between 2 weeks post-intervention change and pre-intervention change (or [(T4-T2)-(T2-T1)]) for the Faith factor of the FACIT-Sp-12
Statistical Analysis 7: Comparison: Writing; Test type: Other; p = .55, Mixed Models Analysis — The above p value refers to the difference between post-intervention change and pre-intervention change (or [(T3-T2)-(T2-T1)]) for the revised Faith factor of the FACIT-Sp-12; Mean Difference (Net) = -0.4 — The above value represents net difference between post-intervention change and pre-intervention change (or [(T3-T2)-(T2-T1)]) for the revised Faith factor of the FACIT-Sp-12
Statistical Analysis 8: Comparison: Writing; Test type: Other; p = .80, Mixed Models Analysis — The above p value refers to the difference between 2 weeks post-intervention change and pre-intervention change (or [(T4-T2)-(T2-T1)]) for the revised Faith factor of the FACIT-Sp-12; Mean Difference (Net) = -0.9 — The above value represents net difference between 2 weeks post-intervention change and pre-intervention change (or [(T4-T2)-(T2-T1)]) for the revised Faith factor of the FACIT-Sp-12
Statistical Analysis 9: Comparison: Writing; Test type: Other; p = .34, Mixed Models Analysis — The above p value refers to the difference between post-intervention change and pre-intervention change (or [(T3-T2)-(T2-T1)]) for the total FACIT-Sp-12 (revised); Mean Difference (Net) = -1.5 — The above value represents net difference between post-intervention change and pre-intervention change (or [(T3-T2)-(T2-T1)]) for the total FACIT-Sp-12 (revised)
Statistical Analysis 10: Comparison: Writing; Test type: Other; p = .91, Mixed Models Analysis — The above p value refers to the difference between 2 weeks post-intervention change and pre-intervention change (or [(T4-T2)-(T2-T1)]) for the total FACIT-Sp-12 (revised); Mean Difference (Net) = -3.0 — The above value represents net difference between 2 weeks post-intervention change and pre-intervention change (or [(T4-T2)-(T2-T1)]) for the total FACIT-Sp-12 (revised)

4. Secondary Outcome: Mean Changes From Baseline in Anxiety and Depression Scores on the Hospital Anxiety and Depression Scale (HADS) to Two-, Six-, and Eight Weeks Post Baseline
Description: Changes include raw score changes and standardized mean differences. Scores on the Hospital Anxiety and Depression Scale (HADS) range from 0 to 42, with higher score indicating higher level of anxiety or depression. The two subscales HADS anxiety (HADS-A) and HADS depression (HADS-D) were analyzed separately. Each sub-scale has a range from 0-21, with the higher score indicating higher level of anxiety or depression.
Time Frame: Baseline (T1) as well as 2 weeks (T2), 6 weeks (T3), and 8 weeks post baseline (T4)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Writing
Number analyzed (Participants) | 54
score on a scale
  HADS-A at T1 | 6.6 (3.9)
  HADS-A at T2 | 5.4 (3.3)
  HADS-A at T3 | 5.7 (4.0)
  HADS-A at T4 | 5.3 (4.1)
  HADS-D at T1 | 4.7 (3.2)
  HADS-D at T2 | 3.9 (2.8)
  HADS-D at T3 | 4.2 (3.5)
  HADS-D at T4 | 4.5 (3.7)
Statistical Analysis 1: Comparison: Writing; We analyzed short- (at 6 weeks post-baseline, T3) and longer-term differences (at 8 weeks post-baseline, T4) for two subscales HADS-A and HADS-D respectively, expecting a larger size of differences at T3. The short-term difference [(T3-T2)-(T2-T1)] represents differences between post-intervention change (T3-T2) and pre-intervention change (T2-T1). Longer-term difference [(T4-T2)-(T2-T1)] represents differences between 2 weeks post-intervention change (T4-T2) and pre-intervention change (T2-T1); Test type: Other; p = .14, Mixed Models Analysis — The above p value refers to the difference between post-intervention change and pre-intervention change (or [(T3-T2)-(T2-T1)]) for HADS-anxiety subscale (HADS-A); Mean Difference (Net) = 1.1 — The above value represents net difference between post-intervention change and pre-intervention change (or [(T3-T2)-(T2-T1)]) for HADS-anxiety subscale (HADS-A)
Statistical Analysis 2: Comparison: Writing; Test type: Other; p = .14, Mixed Models Analysis — The above p value refers to the difference between 2 weeks post-intervention change and pre-intervention change (or [(T4-T2)-(T2-T1)]) for HADS-anxiety subscale (HADS-A); Mean Difference (Net) = 1.2 — The above value represents net difference between 2 weeks post-intervention change and pre-intervention change (or [(T4-T2)-(T2-T1)]) for HADS-anxiety subscale (HADS-A)
Statistical Analysis 3: Comparison: Writing; Test type: Other; p = .32, Mixed Models Analysis — The above p value refers to the difference between post-intervention change and pre-intervention change (or [(T3-T2)-(T2-T1)]) for HADS-depression subscale (HADS-D); Median Difference (Net) = 0.6 — The above value represents net difference between post-intervention change and pre-intervention change (or [(T3-T2)-(T2-T1)]) for HADS-depression subscale (HADS-D)
Statistical Analysis 4: Comparison: Writing; Test type: Other; p = .20, Mixed Models Analysis — The above p value refers to the difference between 2 weeks post-intervention change and pre-intervention change (or [(T4-T2)-(T2-T1)]) for HADS-depression subscale (HADS-D); Mean Difference (Net) = 0.9 — The above value represents net difference between 2 weeks post-intervention change and pre-intervention change (or [(T4-T2)-(T2-T1)]) for HADS-depression subscale (HADS-D)

ADVERSE EVENTS:
Time Frame: Eight weeks following baseline data collection.
Arm/Group | Writing
All-Cause Mortality (participants affected / at risk) | 3/57
Serious Adverse Events (participants affected / at risk) | 0/57
Other Adverse Events (participants affected / at risk) | 0/57

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-03-27): https://cdn.clinicaltrials.gov/large-docs/50/NCT05235750/Prot_SAP_000.pdf